CLINICAL TRIAL: NCT02927366
Title: A Randomized, Parallel-group, Placebo-controlled Subject and Investigator Blinded Study to Assess the Safety, Tolerability, Pharmacokinetics and Efficacy of QCC374 in the Treatment of Pulmonary Arterial Hypertension
Brief Title: Safety, Pharmacokinetics and Efficacy Study of QCC374 in PAH Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated early for strategic reasons. Only Part I of the study was completed.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQCC374X2201; 2016-001412-38 (EudraCT Number)
Record Dates: First submitted 2016-10-05; First posted 2016-10-07 (Estimated); Results first posted 2019-08-07 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-02

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary hypertension (PH),; Increase blood pressure in the pulmonary artery; Increased blood pressure in the pulmonary vein; Increased blood pressure in the lung vasculature; Shortness of breath; Dizziness; Fainting; Leg swelling; Cough; QCC374
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary; Dyspnea; Dizziness; Syncope; Cough

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- QCC374 (Experimental): Adult patients with pulmonary arterial hypertension (PAH) on QCC374. All patients were initiated at 0.03 mg BID (Day 1-3), and were up-titrated to next higher dose 0.06 mg BID (Day 4) and increased to 0.12 mg BID (Day 7-14).
  Interventions: Drug: QCC374
- Placebo (Placebo Comparator): Adult patients with pulmonary arterial hypertension (PAH) on placebo matching to QCC374 doses (0.03 mg BID (Day 1-3), 0.06 mg BID (Day 4) and 0.12 mg BID (Day 7-14)).
  Interventions: Drug: Placebo Matching

INTERVENTIONS:
Drug: QCC374 — 0.03 mg (2 capsules of 0.015 mg) BID 0.06 mg (1 capsule of 0.06 mg) BID 0.12 mg (2 capsules of 0.06 mg) BID
  Arms: QCC374
Drug: Placebo Matching — Placebo matching to QCC374:
  0.03 mg BID, 0.06 mg BID and 0.12 mg BID
  Arms: Placebo

SUMMARY:
This was a non-confirmatory, randomized, placebo controlled, subject and investigator blinded study of QCC374 in PAH subjects. The study was planned to have 2 Parts: Part 1, an initial safety cohort with a 0.03 mg bid starting dose, and Part 2, a larger cohort with a 0.06 mg bid starting dose. However, due to early study termination following Part 1, Part 2 was not completed. Both study parts were comprised of four phases: a screening period for up to 28 days, a titration period of 2 weeks, a stable dose period of 14 weeks and safety follow-up period for 28 days. At the end of the treatment period of 16 weeks, eligible patients were given the option to participate in a separate long-term extension study (CQCC374X2201E1 (NCT02939599)), where all patients were treated with an individual optimal dose of QCC374.

DETAILED DESCRIPTION:
The decision for early termination was based on changes in Novartis strategy, and was not based on any safety concerns regarding QCC374. Only Part 1 of the study was completed.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 years of age or older with symptomatic PAH.
* Subjects with PAH belonging to one of the following subgroups of the Updated Clinical Classification Group 1 (Nice, 2013):
* Idiopathic PAH
* familial PAH
* PAH associated with connective tissue disease, congenital heart disease (surgically repaired at least 12 months prior to screening) or drug or toxin induced (for example, anorexigen use).
* Subjects must have persistent symptoms due to PAH despite therapy with at least one of the following PAH medications: an endothelin receptor antagonist, asoluble guanylate cyclase stimulator or a phosphodiesterase inhibitor. The subjects' PAH medication regimen, with typical medications including calcium channel blockers, endothelin receptor antagonists, soluble guanylate cyclase stimulators and/or phosphodiesterase inhibitors, must have been used at a stable dose and frequency for at least 12 weeks before the screening visit and during the screening period.
* Diagnosis of PAH established according to the standard criteria before the screening visit:
* Resting mean pulmonary arterial pressure > 25 mmHg.
* PVR > 240 dynes s/cm5.
* Pulmonary capillary wedge pressure or left ventricular end diastolic pressure < 15 mmHg
* PVR > 400 dynes s/cm5 at the time of the baseline right heart catheterization (RHC) (if a RHC was completed within one month of the screening visit, that result may be used for inclusion).
* 6-minute walk distance greater than 150 meters at Screening. This distance must be confirmed by a second 6MWT prior to randomization. The value of the second 6MWD should be within ± 15% of the value obtained at Screening.

Exclusion Criteria:

* Subjects with clinically unstable right heart failure within the last three months (New York Heart Association (NYHA) Class IV).
* Subjects with PAH associated with portal hypertension, Human Immunodeficiency Virus (HIV) infection or unrepaired congenital systemic to pulmonary shunts
* Subjects who have received or have been scheduled to receive long-term treatment with epoprostenol or any prostacyclin within the three months prior to the screening visit or during the screening period.
* Hypotensive subjects (systemic systolic blood pressure < 85 mmHg)
* Subjects with a history of left sided heart disease, chronic left sided heart failure, congenital or acquired valvular disease and/or pulmonary venous hypertension.
* Subjects with significant obstructive (forced expiratory volume in one second [FEV1]/forced vital capacity [FVC] < 70% predicted) or restrictive (total lung capacity < 70% predicted) lung disease at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- Novartis Investigative Site, Pittsburgh, Pennsylvania, United States
- Germany (2):
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Heidelberg
- Novartis Investigative Site, Seoul, South Korea
- Novartis Investigative Site, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=403

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 5 centers in 4 countries: Germany (2), Korea (1), UK (1) and USA (1).
Pre-assignment Details: Part 1 consisted of 8 subjects, randomized in a 6:2 ratio to QCC374 or placebo. The planned bid dose levels in Part 1 were 0.03 mg, 0.06 mg and 0.12 mg. Subjects began dosing at 0.03 mg bid.
Period: Overall Study
Arm/Group | QCC374 | Placebo
Started (All randomized patients were included in the Safety Analysis Set (SAF).) | 6 | 2
Pharmacodynamic (PD) Analysis Set (At least one dose of study drug and one evaluable PD assessment) | 6 | 2
Pharmacokinetic (PK) Analysis Set (At least one dose of study drug and one evaluable PK concentration measurement) | 4 | 0
Completed | 4 | 2
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Patient schedule | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QCC374 | Placebo | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.0 (14.62) | 57.5 (9.19) | 45.1 (14.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 0 | 1
  White | 5 | 2 | 7
Ethiology of Pulmonary Arterial Hypertension (PAH) [Count of Participants; unit: Participants]
  Family PAH | 1 | 0 | 1
  Idiopathic PAH | 4 | 1 | 5
  PAH associated with Connective Tissue Disease | 1 | 0 | 1
  PAH induced by Drug/Toxin | 0 | 1 | 1
Time from Pulmonary Arterial Hypertension (PAH) diagnosis [Median (Full Range); unit: Years] | 2.985 [0.56 to 7.77] | 9.201 [6.04 to 12.36] | 4.966 [0.56 to 12.36]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pulmonary Vascular Resistance (PVR) at Week 16 (Day 111)
Description: The efficacy of 16 weeks of QCC374 administration in subjects with Pulmonary Arterial Hypertension (PAH) was assessed by measuring changes from baseline in Pulmonary Vascular Resistance (PVR). PVR is derived from the CO measurement in dyn·s/cm5 and can be calculated as 80 multiplied by (Mean Arterial Pressure - Mean Pulmonary Artery Wedge Pressure) divided by Cardiac Output. A higher negative number in Pulmonary Vascular Resistance indicates improvement. Only descriptive analysis performed.
Time Frame: Baseline, Week 16 (Day 111)
Population: Participants from the Pharmacodynamic (PD) analysis set, defined as all randomized participants who received at least one dose of study drug and one evaluable PD assessment, with data available for analysis were considered.
Measure: Mean (Standard Deviation); unit: dyn*s/cm5
Arm/Group | QCC374 | Placebo
Number analyzed (Participants) | 6 | 2
dyn*s/cm5
  PVR at Screening-Ratio to Baseline | 1.00 (0.000) | 1.00 (0.000)
  PVR at Day 111-Ratio to Baseline: number analyzed (Participants) | 4 | 2
  PVR at Day 111-Ratio to Baseline | 1.07 (0.274) | 1.05 (0.073)

2. Secondary Outcome: Change From Baseline in Six Minute Walk Distance (6MWD) Over Time
Description: The Six Minute Walk Test measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is able to self-pace and rest as needed as they traverse back and forth along a marked walkway. Only descriptive analysis performed.
Time Frame: Baseline, Day 28, Day 56, Day 84 and Day 111
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Meter
Arm/Group | QCC374 | Placebo
Number analyzed (Participants) | 6 | 2
Meter
  Baseline | 443.83 (47.942) | 458.50 (111.723)
  Chge from BL at Day 28 | -7.17 (20.651) | 9.75 (13.789)
  Chge from BL at Day 56: number analyzed (Participants) | 5 | 2
  Chge from BL at Day 56 | -11.60 (19.562) | 14.50 (19.799)
  Chge from BL at Day 84: number analyzed (Participants) | 4 | 2
  Chge from BL at Day 84 | -4.25 (21.956) | 12.50 (16.971)
  Chge from BL at Day 111: number analyzed (Participants) | 4 | 2
  Chge from BL at Day 111 | 13.25 (25.002) | 14.00 (9.192)

3. Secondary Outcome: Change From Baseline in Cardiac Output (CO) at Week 16 (Day 111)
Description: The Right Heart Catheterization (RHC) assessment was performed to assess several hemodynamic variables in pulmonary hypertension, including Cardiac Output (CO). All hemodynamic parameters were assessed when the patient was in a stable hemodynamic rest state (as demonstrated by three consecutive CO measurements within 10% of each other) while the patient was breathing ambient air or oxygen. CO was measured in triplicate using the thermodilution technique. Direct Fick could be used only after discussion and approval by the Sponsor. In all cases, the same technique was to be used at baseline and week 16. . A higher positive number in Cardiac Output indicates improvement. Only descriptive analysis performed.
Time Frame: Baseline, Week 16 (Day 111)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | QCC374 | Placebo
Number analyzed (Participants) | 6 | 2
L/min
  Average Cardiac Output at Baseline | 4.33 (1.527) | 3.61 (0.085)
  Average Cardiac Output at Day 111: number analyzed (Participants) | 4 | 2
  Average Cardiac Output at Day 111 | 4.46 (0.937) | 3.79 (0.191)
  Cardiac Output 1 at Baseline | 4.38 (1.491) | 3.61 (0.127)
  Cardiac Output 1 at Day 111: number analyzed (Participants) | 4 | 2
  Cardiac Output 1 at Day 111 | 4.58 (1.002) | 3.69 (0.311)
  Cardiac Output 2 at Baseline: number analyzed (Participants) | 5 | 2
  Cardiac Output 2 at Baseline | 3.96 (1.588) | 3.60 (0.000)
  Cardiac Output 2 at Day 111: number analyzed (Participants) | 3 | 2
  Cardiac Output 2 at Day 111 | 4.33 (0.993) | 3.89 (0.233)
  Cardiac Output 3 at Baseline: number analyzed (Participants) | 5 | 2
  Cardiac Output 3 at Baseline | 3.98 (1.340) | 3.61 (0.127)
  Cardiac Output 3 at Day 111: number analyzed (Participants) | 3 | 2
  Cardiac Output 3 at Day 111 | 4.40 (1.238) | 3.79 (0.028)

4. Secondary Outcome: Change From Baseline in Cardiac Index at Week 16 (Day 111)
Description: The Right Heart Catheterization (RHC) assessment was performed to assess several hemodynamic variables in pulmonary hypertension, including Cardiac Index. All hemodynamic parameters were assessed when the patient was in a stable hemodynamic rest state (as demonstrated by three consecutive CO measurements within 10% of each other) while the patient was breathing ambient air or oxygen. A higher negative number in Cardiac Index indicates improvement. Only descriptive analysis performed.
Time Frame: Baseline, Week 16 (Day 111)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/min/m2
Arm/Group | QCC374 | Placebo
Number analyzed (Participants) | 6 | 2
L/min/m2
  Cardiac Index at Baseline | 2.45 (0.794) | 2.15 (0.070)
  Cardiac Index at Day 111: number analyzed (Participants) | 1 | 0
  Cardiac Index at Day 111 | 2.54 (NA) — NA: Not estimable due to insufficient number of participants with events |

5. Secondary Outcome: Change From Baseline in Pulmonary Capillary Wedge Pressure (PCWP) at Week 16 (Day 111)
Description: The Right Heart Catheterization (RHC) assessment was performed to assess several hemodynamic variables in pulmonary hypertension, including mean Pulmonary Capillary Wedge Pressure (PCWP). All hemodynamic parameters were assessed when the patient was in a stable hemodynamic rest state (as demonstrated by three consecutive CO measurements within 10% of each other) while the patient was breathing ambient air or oxygen. Pressure measurements were made in the PA, PA wedge, right ventricle (RV) and right atrium (RA) and determined at the end of normal expiration. The PCWP was recorded as the mean of three measurements. Only descriptive analysis performed.
Time Frame: Baseline, Week 16 (Day 111)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | QCC374 | Placebo
Number analyzed (Participants) | 6 | 2
mmHg
  PCWP at Baseline | 8.67 (1.366) | 9.50 (0.707)
  PCWP at Day 111: number analyzed (Participants) | 4 | 2
  PCWP at Day 111 | 11.75 (5.188) | 9.50 (0.707)

6. Secondary Outcome: Change From Baseline in Systemic Vascular Resistance (SVR) at Week 16 (Day 111)
Description: The Right Heart Catheterization (RHC) assessment was performed to assess several hemodynamic variables in pulmonary hypertension, including Systemic Vascular Resistance (SVR). All hemodynamic parameters were assessed when the patient was in a stable hemodynamic rest state (as demonstrated by three consecutive CO measurements within 10% of each other) while the patient was breathing ambient air or oxygen. SVR is derived from the CO measurement in dyn·s/cm5 and can be calculated as 80 multiplied by (Mean Arterial Pressure - Mean Venous Pressure or CVP)) divided by Cardiac Output. A higher negative number in Mean Systemic Vascular Resistance indicates improvement. Only descriptive analysis performed.
Time Frame: Baseline, Week 16 (Day 111)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dynes*Sec*cm5
Arm/Group | QCC374 | Placebo
Number analyzed (Participants) | 6 | 2
dynes*Sec*cm5
  SVR at Baseline: number analyzed (Participants) | 5 | 2
  SVR at Baseline | 1133.31 (410.336) | 1425.89 (633.723)
  SVR at Day 111: number analyzed (Participants) | 2 | 2
  SVR at Day 111 | 1285.50 (465.983) | 1240.00 (274.357)

7. Secondary Outcome: Change From Baseline in RV Fractional Area Change and RV Free Wall Average Peak Long Strain at Week 16 (Day 111) Using Echocardiography
Description: Key Right Ventricular (RV) function endpoints such as RV fractional area change (RV FAC) and RV Free Wall Average Peak Long Strain (RV FWPLS) were assessed with echocardiography. A higher number in RV FAC and a lower number in RV FWPLS indicate an improvement. Only descriptive analysis performed.
Time Frame: Baseline, Week 16 (Day 111)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | QCC374 | Placebo
Number analyzed (Participants) | 5 | 2
Percentage
  RV FAC at Baseline: number analyzed (Participants) | 4 | 2
  RV FAC at Baseline | 20.17 (8.717) | 30.05 (7.050)
  RV FAC at Day 111: number analyzed (Participants) | 2 | 1
  RV FAC at Day 111 | 20.70 (5.091) | 26.20 (NA) — NA: Not estimable due to insufficient number of participants with events
  RV FWPLS at Baseline: number analyzed (Participants) | 5 | 1
  RV FWPLS at Baseline | 12.68 (3.534) | 16.30 (NA) — NA: Not estimable due to insufficient number of participants with events
  RV FWPLS at Day 111: number analyzed (Participants) | 2 | 0
  RV FWPLS at Day 111 | 7.85 (2.758) |

8. Secondary Outcome: Change From Baseline in RV Tei Index at Week 16 (Day 111) Using Echocardiography
Description: Key Right Ventricular (RV) function endpoints such as Tei Index were assessed with echocardiography. The RV Tei index is using both systolic and diastolic time intervals to evaluate the overall global dysfunction of the right ventricle in PAH patients. A lower number in RV Tei Index indicates an improvement. Only descriptive analysis performed.
Time Frame: Baseline, Week 16 (Day 111)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | QCC374 | Placebo
Number analyzed (Participants) | 5 | 2
Index
  RV Tei Index at Baseline: number analyzed (Participants) | 4 | 2
  RV Tei Index at Baseline | 0.92 (0.260) | 0.88 (0.361)
  RV Tei Index at Day 111: number analyzed (Participants) | 2 | 2
  RV Tei Index at Day 111 | 0.89 (0.099) | 0.89 (0.078)

9. Secondary Outcome: Change From Baseline in Tricuspid Annular Peak Systolic Velocity (TA S') at Week 16 (Day 111) Using Echocardiography
Description: Key Right Ventricular (RV) function endpoints such as Tricuspid Annular Peak Systolic Velocity (TA S') were assessed with echocardiography. Only descriptive analysis performed.
Time Frame: Baseline, Week 16 (Day 111)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | QCC374 | Placebo
Number analyzed (Participants) | 5 | 2
cm/s
  TA S' at Baseline: number analyzed (Participants) | 4 | 2
  TA S' at Baseline | 11.23 (1.723) | 9.50 (0.990)
  TA S' at Day 111: number analyzed (Participants) | 3 | 1
  TA S' at Day 111 | 9.73 (1.069) | 13.20 (NA) — NA: Not estimable due to insufficient number of participants with events

10. Secondary Outcome: Change From Baseline in Tricuspid Annular Plane Sys Excursion (TAPSE) at Week 16 (Day 111) Using Echocardiography
Description: Key Right Ventricular (RV) function endpoints such as Tricuspid Annular Plane Sys Excursion (TAPSE) were assessed with echocardiography. A higher number in TAPSE indicates an improvement. Only descriptive analysis performed.
Time Frame: Baseline, Week 16 (Day 111)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | QCC374 | Placebo
Number analyzed (Participants) | 5 | 2
cm
  TAPSE at Baseline: number analyzed (Participants) | 4 | 2
  TAPSE at Baseline | 1.88 (0.313) | 1.27 (0.170)
  TAPSE at Day 111: number analyzed (Participants) | 3 | 1
  TAPSE at Day 111 | 1.79 (0.511) | 1.76 (NA) — NA: Not estimable due to insufficient number of participants with events

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for QCC374 and Its Metabolite QCM441
Description: Cmax is the maximum (peak) observed plasma drug concentration after single dose administration. PK parameters were calculated from plasma concentration-time data using non-compartmental methods. Only descriptive analysis performed.
Time Frame: Day 1 and 112 (0.00, 0.05, 0.15, 0.30, 1.00, 2.00, 4.00, 8.00 and 12.00 hours post-dose))
Population: Participants from the Pharmacokinetic (PK) analysis set, defined as all randomized participants who received at least one dose of study drug and one evaluable PK concentration measurement, with data available for analysis were considered.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | QCC374 | Placebo
Number analyzed (Participants) | 4 | 0
pg/mL
  QCC374: Day 1, Dose Level 0.03 mg | 101 (15.7) |
  QCC374: Day 112, Dose Level 0.06 mg: number analyzed (Participants) | 1 | 0
  QCC374: Day 112, Dose Level 0.06 mg | 461 (NA) — NA: Not estimable due to insufficient number of participants with events |
  QCC374: Day 112, Dose Level 0.12 mg: number analyzed (Participants) | 1 | 0
  QCC374: Day 112, Dose Level 0.12 mg | 406 (NA) — NA: Not estimable due to insufficient number of participants with events |
  QCM441: Day 1, Dose Level 0.03 mg | 346 (32.4) |
  QCM441: Day 112, Dose Level 0.06 mg: number analyzed (Participants) | 1 | 0
  QCM441: Day 112, Dose Level 0.06 mg | 2350 (NA) — NA: Not estimable due to insufficient number of participants with events |
  QCM441: Day 112, Dose Level 0.12 mg: number analyzed (Participants) | 1 | 0
  QCM441: Day 112, Dose Level 0.12 mg | 3610 (NA) — NA: Not estimable due to insufficient number of participants with events |

12. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) for QCC374 and Its Metabolite QCM441
Description: Tmax is the time to reach maximum plasma concentration after single dose administration. PK parameters were calculated from plasma concentration-time data using non-compartmental methods. Only descriptive analysis performed.
Time Frame: Day 1 and 112 (0.00, 0.05, 0.15, 0.30, 1.00, 2.00, 4.00, 8.00 and 12.00 hours post-dose))
Population: as for outcome 11
Measure: Median (Full Range); unit: hour
Arm/Group | QCC374 | Placebo
Number analyzed (Participants) | 4 | 0
hour
  QCC374: Day 1, Dose Level 0.03 mg | 0.159 [0.0830 to 0.267] |
  QCC374: Day 112, Dose Level 0.06 mg: number analyzed (Participants) | 1 | 0
  QCC374: Day 112, Dose Level 0.06 mg | 0.00 [0.00 to 0.00] |
  QCC374: Day 112, Dose Level 0.12 mg: number analyzed (Participants) | 1 | 0
  QCC374: Day 112, Dose Level 0.12 mg | 0.517 [0.517 to 0.517] |
  QCM441: Day 1, Dose Level 0.03 mg | 3.99 [3.85 to 8.00] |
  QCM441: Day 112, Dose Level 0.06 mg: number analyzed (Participants) | 1 | 0
  QCM441: Day 112, Dose Level 0.06 mg | 1.00 [1.00 to 1.00] |
  QCM441: Day 112, Dose Level 0.12 mg: number analyzed (Participants) | 1 | 0
  QCM441: Day 112, Dose Level 0.12 mg | 4.02 [4.02 to 4.02] |

13. Secondary Outcome: Area Under the Plasma Concentration-time Curve From 0 to the Last Measurable Concentration (AUClast) for QCC374 and Its Metabolite QCM441
Description: AUClast is the area under the plasma concentration-time curve from time zero to the last measurable concentration sampling time. PK parameters were calculated from plasma concentration-time data using non-compartmental methods. Only descriptive analysis performed.
Time Frame: Day 1 and 112 (0.00, 0.05, 0.15, 0.30, 1.00, 2.00, 4.00, 8.00 and 12.00 hours post-dose))
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | QCC374 | Placebo
Number analyzed (Participants) | 4 | 0
h*pg/mL
  QCC374: Day 1, Dose Level 0.03 mg | 128 (14.3) |
  QCC374: Day 112, Dose Level 0.06 mg: number analyzed (Participants) | 1 | 0
  QCC374: Day 112, Dose Level 0.06 mg | 638 (NA) — NA: Not estimable due to insufficient number of participants with events |
  QCC374: Day 112, Dose Level 0.12 mg: number analyzed (Participants) | 1 | 0
  QCC374: Day 112, Dose Level 0.12 mg | 883 (NA) — NA: Not estimable due to insufficient number of participants with events |
  QCM441: Day 1, Dose Level 0.03 mg | 2590 (22.8) |
  QCM441: Day 112, Dose Level 0.06 mg: number analyzed (Participants) | 1 | 0
  QCM441: Day 112, Dose Level 0.06 mg | 17700 (NA) — NA: Not estimable due to insufficient number of participants with events |
  QCM441: Day 112, Dose Level 0.12 mg: number analyzed (Participants) | 1 | 0
  QCM441: Day 112, Dose Level 0.12 mg | 33800 (NA) — NA: Not estimable due to insufficient number of participants with events |

14. Secondary Outcome: Area Under the Plasma Concentration Time Curve From 0 to the End of a Dosing Interval (AUCtau) for QCC374 and Its Metabolite QCM441
Description: AUCtau is the area under the plasma concentration-time curve from time zero to the end of the dosing interval. PK parameters were calculated from plasma concentration-time data using non-compartmental methods. Only descriptive analysis performed.
Time Frame: Day 1 and 112 (0.00, 0.05, 0.15, 0.30, 1.00, 2.00, 4.00, 8.00 and 12.00 hours post-dose))
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | QCC374 | Placebo
Number analyzed (Participants) | 4 | 0
h*pg/mL
  QCC374: Day 1, Dose Level 0.03 mg | 148 (15.5) |
  QCC374: Day 112, Dose Level 0.06 mg: number analyzed (Participants) | 1 | 0
  QCC374: Day 112, Dose Level 0.06 mg | 638 (NA) — NA: Not estimable due to insufficient number of participants with events |
  QCC374: Day 112, Dose Level 0.12 mg: number analyzed (Participants) | 1 | 0
  QCC374: Day 112, Dose Level 0.12 mg | 910 (NA) — NA: Not estimable due to insufficient number of participants with events |
  QCM441: Day 1, Dose Level 0.03 mg | 2600 (40.6) |
  QCM441: Day 112, Dose Level 0.06 mg: number analyzed (Participants) | 1 | 0
  QCM441: Day 112, Dose Level 0.06 mg | 17700 (NA) — NA: Not estimable due to insufficient number of participants with events |
  QCM441: Day 112, Dose Level 0.12 mg: number analyzed (Participants) | 1 | 0
  QCM441: Day 112, Dose Level 0.12 mg | 33800 (NA) — NA: Not estimable due to insufficient number of participants with events |

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events were collected for the maximum duration of participants' treatment exposure plus any follow up period, approximately 5 months.
Arm/Group | QCC374 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/2
Other Adverse Events (participants affected / at risk) | 6/6 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QCC374 (N=6) | Placebo (N=2)
Syncope (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QCC374 (N=6) | Placebo (N=2)
Dental Caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Disorder (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Hangover (General disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1
Otitis Media (Infections and infestations) | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Head Discomfort (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 5 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 3 | 0

LIMITATIONS AND CAVEATS:
Due to the limited number of subjects with the available data at Week 16 (Day 111), for the primary and secondary efficacy endpoints, it is not possible to draw any meaningful treatment comparisons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/66/NCT02927366/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT02927366/SAP_001.pdf